CLINICAL TRIAL: NCT01550224
Title: Temozolomide Plus Vorinostat in Patients With Relapse/Refractory Acute Myeloid Leukemia (AML)
Brief Title: Temozolomide Plus Vorinostat in Relapse/Refractory Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steven E. Coutre (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Steven E. Coutre, Professor of Medicine (Hematology), Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-22794; NCT01550224 (Other: Stanford University); HEMAML0017 (Other: OnCore)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Acute Myeloid Leukemia With 11q23-abnormality in Relapse
MeSH Terms: interventions — Temozolomide; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participant Group 1 (methylated MGMT promoter) (Active Comparator): Participants with methylated O6-methylguanine DNA methyltransferase (MGMT) promoter, ie, expected to have no expression of MGMT protein, will be assigned into Group 1, and will receive vorinostat 500 mg orally 3 times daily for 3 days, followed by conventional doses of temozolomide (200 mg/m2 for 7 days).
  Interventions: Drug: Temozolomide; Drug: Vorinostat
- Participant Group 2 (non-methylated MGMT promoter) (Active Comparator): Participants with non-methylated O6-methylguanine DNA methyltransferase (MGMT) promoter, ie, expected to have expression MGMT protein, will be assigned to into Group 2, and will initially receive daily, low doses (protracted dose schedule) of temozolomide (100 mg/m2) for 14 days in an attempt to inactivate MGMT activity. Following the protracted dose schedule, participants will receive vorinostat 500 mg orally 3 times daily for 3 days, followed by conventional doses of temozolomide (200 mg/m2 for 7 days).
  Interventions: Drug: Temozolomide; Drug: Vorinostat

INTERVENTIONS:
Drug: Temozolomide — An alkylating agent administered for induction per standard of care at 200 mg/m²/day for 7days.
  Other Names: Temodar; Temodal; Temcad; TMZ
Drug: Vorinostat — A synthetic hydroxamic acid derivative with antineoplastic activity administered for both groups at 500 mg orally 3 times daily for 3 days prior to Temozolomide 200 mg/m²/day.
  Other Names: Zolinza

SUMMARY:
The purpose of the study is to first determine if temozolomide plus vorinostat in combination can control relapsed or refractory acute myeloid leukemia (AML) and determine if this combination can be safely taken. The study will look at the side effects of the Temozolomide plus Vorinostat in combination and whether the treatment schedule is tolerated.

DETAILED DESCRIPTION:
The primary endpoint of the study is to determine the clinical efficacy as determined by the rate of morphological complete remission, of 2 different treatment regimens of temozolomide and vorinostat administered to 2 distinct groups of participants patients with AML and poor prognostic features. Participants will be allocated to treatment on the basis of O6-methylguanine DNA methyltransferase (MGMT) promoter methylation status.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically- or cytologically-confirmed acute myeloid leukemia (AML)
* Relapsed or refractory (AML), after at least 1 prior induction regimen
* Age ≥ 18 years
* Life expectancy > 2 months.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Calculated creatinine clearance ≤ 2.0 mg/dL (OR ≥ 30 mL/min for patients with serum creatinine levels > 2.0 mg/dL)
* Serum total bilirubin ≤ 1.5 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 X ULN
* Alanine aminotransferase (ALT) ≤ 2.5 X ULN
* Alkaline phosphatase (liver fraction) ≤ 2.5 X ULN
* If male, must agree to use an adequate method of contraception for the duration of the study and 1 month following coming off study or of study completion
* If female of childbearing potential, must a negative serum pregnancy test within 72 hours prior to receiving the first dose of vorinostat.
* If female, must be one of the following:

  * Post-menopausal (free from menses for ≥ 2 years),
  * Surgically-sterilized
  * Willing to use 2 adequate barrier methods of contraception
  * Agree to abstain from heterosexual activity throughout the study, starting with Visit 1
* Available at the treating institution for study assessments and procedures for the duration of the study
* Written informed consent

EXCLUSION CRITERIA

* Received chemotherapy; radiotherapy; or biological therapy within 30 days (42 days for nitrosoureas or mitomycin C) prior to initial dosing with study drug(s), or has not recovered from adverse events due to agents administered more than 30 days earlier, except for hydroxyurea-related adverse events.
* Currently participating or within 30 days of initial dosing with study drug(s), has participated in a study with an investigational compound or device
* Receiving any other investigational agents or concomitant radiotherapy, chemotherapy, or immunotherapy.
* Received a histone deacetylase (HDAC) inhibitor [eg, romidepsin (Depsipeptide), NSC-630176, MS 275, LAQ-824, belinostat (PXD-101), LBH589, MGCD0103, CRA024781, etc] within the past 30 days. Patients who have received valproic acid or other compounds with HDAC inhibitor-like activity, as anti-tumor therapy should not enroll in this study. Patients who have received such compounds for other indications, eg, valproic acid for epilepsy, may enroll after a 30-day washout period.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide; vorinostat; dacarbazine (DTIC-Dome, DIC, imidazole carboxamide)
* History of gastrointestinal disease or significant bowel resection that could interfere with drug absorption or inability to swallow tablets.
* Uncontrolled intercurrent illness (as defined by the investigators) including, but not limited to, ongoing or active infection (HIV, Hepatitis B or Hepatitis C), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Prior allogeneic stem cell transplantation within 2 months of trial enrollment or prior radiation up to more than 25% of bone marrow.
* Currently active 2nd malignancy, other than nonmelanoma skin cancer and carcinoma in situ of the cervix (completed therapy for a prior malignancy, and disease-free from prior malignancies for >5 years or are considered by their physician to be at less than 30% risk of relapse is not considered to be an "currently active" malignancy)
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnant or breast feeding
* Expecting to conceive or father children within the projected duration of the study.
* Uncontrolled intercurrent illness or circumstances that could limit compliance with the study, including, but not limited to the following: active infection, acute or chronic graft versus host disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric conditions.
* History or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2014-11-17 (Actual); Study Completion 2014-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Coutre, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participant Group 1 (Methylated MGMT Promoter): Participants with methylated O6-methylguanine DNA methyltransferase (MGMT) promoter, ie, expected to have no expression of MGMT protein, will be assigned into Group 1, and will receive vorinostat 500 mg orally 3 times daily for 3 days, followed by conventional doses of temozolomide (200 mg/m2 for 7 days).
  Temozolomide: An alkylating agent administered for induction per standard of care at 200 mg/m²/day for 7days. Group 2 participants also receive at protracted, pre-induction treatment with 100 mg/m²/day for 14 days.
  Vorinostat: A synthetic hydroxamic acid derivative with antineoplastic activity administered for both groups at 500 mg orally 3 times daily for 3 days prior to Temozolomide 200 mg/m²/day.
Period: Overall Study
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter)
Started | 3 | 20
Completed | 3 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter) | Total
Number analyzed (Participants) | 3 | 20 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 3 | 20 | 23
Age, Continuous [Median (Full Range); unit: years] | 76.3 [71 to 85] | 83 [72.4 to 89.3] | 82.7 [71 to 89.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 1 | 15 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 17 | 20
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 15 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 20 | 23

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR)
Description: This study evaluates the clinical efficacy of temozolomide + vorinostat as administered to Groups 1 and 2, assessed as the rate of complete remission [CR, aka morphologic complete remission (mCR)], defined as the morphologic leukemia-free state (MLFS), WITH absolute neutrophil count (ANC) ≥ 1,000/µL AND platelets (PLT) ≥ 100,000/µL. The outcome is reported as the percentage without dispersion of participants in Groups 1 and 2 that demonstrated CR. CR is defined as all of the following.
  MLFS = < 5% blasts in bone marrow aspirate containing marrow spicules > 200 nucleated cells no blasts with Auer rods no persistence of extramedullary disease ANC = ≥ 1,000/µL PLT = ≥ 100,000/µL
Time Frame: up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter)
Number analyzed (Participants) | 3 | 20
Participants | 0 | 0

2. Secondary Outcome: Morphologic Leukemia-free State (MLFS)
Description: The rate of morphologic leukemia-free state (MLFS) is reported as the percentage without dispersion of participants in Groups 1 and 2 that achieve MLFS. The outcome is reported as the percentage without dispersion of participants in Groups 1 and 2 that demonstrated MLFS. This assessment is independent of absolute neutrophil count (ANC) or platelets (PLT) recovery status. MLFS is defined below.
  MLFS = < 5% blasts in bone marrow aspirate containing marrow spicules > 200 nucleated cells no blasts with Auer rods no persistence of extramedullary disease
Time Frame: up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter)
Number analyzed (Participants) | 3 | 20
Participants | 0 | 1

3. Secondary Outcome: Complete Remission With Incomplete Blood Count Recovery (CRp)
Description: The rate of complete remission with incomplete blood count recovery (CRp) for Groups 1 and 2 was assessed as the rate of morphologic leukemia-free state (MLFS) but with EITHER residual neutropenia (ANC < 1,000/µL) OR residual thrombocytopenia (PLT < 100,000/µL). MLFS is defined as follows.
  MLFS = < 5% blasts in bone marrow aspirate containing marrow spicules > 200 nucleated cells no blasts with Auer rods no persistence of extramedullary disease
Time Frame: up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter)
Number analyzed (Participants) | 3 | 20
Participants | 0 | 1

4. Secondary Outcome: Cytogenetic Response (CyR)
Description: Cytogenetic response (CyR) is defined as complete remission (CR), PLUS a documented decrease or absence of cytogenetic abnormalities, when analyzed microscopically for 20 cellular metaphases (actively dividing cells). The outcome is reported as the percentage without dispersion of participants in Groups 1 and 2 that demonstrated CyR. CR is defined as all of the following.
  CR = < 5% blasts in bone marrow aspirate containing marrow spicules; > 200 nucleated cells no blasts with Auer rods; no persistence of extramedullary disease absolute neutrophil count (ANC) ≥ 1,000/µL platelets (PLT) ≥ 100,000/µL
Time Frame: up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter)
Number analyzed (Participants) | 3 | 20
Participants | 0 | 0

5. Secondary Outcome: Partial Remission (PR)
Description: Partial remission (PR) is reported as the percentage without dispersion of participants in Groups 1 and 2 that demonstrated PR. PR is defined as all of the following.
  PR = 5% to 25% blasts (must be ≥ 50% reduction of blasts) in bone marrow aspirate containing marrow spicules; > 200 nucleated cells no blasts with Auer rods no persistence of extramedullary disease absolute neutrophil count (ANC) ≥ 1,000/µL platelets (PLT) ≥ 100,000/µL
Time Frame: up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter)
Number analyzed (Participants) | 3 | 20
Participants | 0 | 0

6. Secondary Outcome: Treatment Failure (TF)
Description: Treatment failure (TF) is defined as failing to achieve either a complete remission (CR) or partial remission (PR) after induction chemotherapy. The outcome is reported as the percentage without dispersion of participants in Groups 1 and 2 that experienced TF. CR and PR are defined as the following.
  CR = < 5% blasts in bone marrow aspirate containing marrow spicules; > 200 nucleated cells no blasts with Auer rods; no persistence of extramedullary disease absolute neutrophil count (ANC) ≥ 1,000/µL platelets (PLT) ≥ 100,000/µL
  PR = 5% to 25% blasts (must be ≥ 50% reduction of blasts) in bone marrow aspirate containing marrow spicules; > 200 nucleated cells no blasts with Auer rods no persistence of extramedullary disease absolute neutrophil count (ANC) ≥ 1,000/µL platelets (PLT) ≥ 100,000/µL
Time Frame: up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter)
Number analyzed (Participants) | 3 | 20
Participants | 3 | 20

7. Secondary Outcome: Disease-free Survival (DFS) at 2 Years
Description: Disease-Free Survival (DFS) is defined as survival after complete response (CR) without disease progression. DFS is reported as the percentage without dispersion of participants in Groups 1 and 2 that experienced CR and were alive without progression (ie, without disease) 2 years after induction chemotherapy. CR is defined as all of the following.
  CR = < 5% blasts in bone marrow aspirate containing marrow spicules; > 200 nucleated cells no blasts with Auer rods; no persistence of extramedullary disease absolute neutrophil count (ANC) ≥ 1,000/µL platelets (PLT) ≥ 100,000/µL
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter)
Number analyzed (Participants) | 3 | 20
Participants | 0 | 0

8. Secondary Outcome: Relapse-Free Survival (RFS) at 2 Years
Description: Relapse-free survival (RFS) is defined as survival after complete response (CR) or (PR) without further disease progression. RFS is reported as the percentage without dispersion of participants in Groups 1 and 2 that experienced CR or PR, and were alive without progression 2 years after induction chemotherapy. CR and PR are defined as the following.
  CR = < 5% blasts in bone marrow aspirate containing marrow spicules; > 200 nucleated cells no blasts with Auer rods; no persistence of extramedullary disease absolute neutrophil count (ANC) ≥ 1,000/µL platelets (PLT) ≥ 100,000/µL
  PR = 5% to 25% blasts (must be ≥ 50% reduction of blasts) in bone marrow aspirate containing marrow spicules; > 200 nucleated cells no blasts with Auer rods no persistence of extramedullary disease absolute neutrophil count (ANC) ≥ 1,000/µL platelets (PLT) ≥ 100,000/µL
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter)
Number analyzed (Participants) | 3 | 20
Participants | 0 | 0

9. Secondary Outcome: Overall Survival (OS) at 2 Years
Description: Overall Survival (OS) is defined as survival regardless of clinical status. OS is reported as the percentage without dispersion of participants in Groups 1 and 2 that remained alive 2 years after induction chemotherapy.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter)
Number analyzed (Participants) | 3 | 20
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Participant Group 1 (Methylated MGMT Promoter) | Participant Group 2 (Non-methylated MGMT Promoter)
All-Cause Mortality (participants affected / at risk) | 3/3 | 20/20
Serious Adverse Events (participants affected / at risk) | 0/3 | 11/20
Other Adverse Events (participants affected / at risk) | 3/3 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participant Group 1 (Methylated MGMT Promoter) (N=3) | Participant Group 2 (Non-methylated MGMT Promoter) (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Hemorrhage (bleeding), subdural hematoma (Vascular disorders) | 0 (0) | 1 (1)
Infection - E coli bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Infection - neutropenic fever (Infections and infestations) | 0 (0) | 4 (4)
Infection - pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Infection - Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Thrombocytopenia (platelet count decreased) (Investigations) | 0 (0) | 1 (1)
Pulmonary/Upper Respiratory - Hemoptysis (coughing up blood) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participant Group 1 (Methylated MGMT Promoter) (N=3) | Participant Group 2 (Non-methylated MGMT Promoter) (N=20)
Anemia (reduced level of red blood cells) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (reduced level of white blood cells) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Low hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (reduced level of neutrophils) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenic fever (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (reduced level of many or all blood cells) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (reduced level of platlets) (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Arrhythmia (irregular heart beat) (Cardiac disorders) | 0 (0) | 2 (2)
Hypotension (low blood pressure) (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal or epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Gastrointestinal disorders) | 0 (0) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 9 (9)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Loss of appetite (Gastrointestinal disorders) | 2 (2) | 1 (1)
Melena (blood in stool) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8)
Rectal abscess (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 7 (7)
Back pain (General disorders) | 0 (0) | 1 (1)
Dysgeusia (altered sense of taste) (General disorders) | 0 (0) | 2 (2)
Elevated serum lactase (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 10 (10)
Limb edema (swelling in extremities) (General disorders) | 0 (0) | 3 (3)
Maceration (General disorders) | 0 (0) | 1 (1)
Night sweat (General disorders) | 0 (0) | 1 (1)
Skin infection (boil) (General disorders) | 0 (0) | 1 (1)
Weakness (General disorders) | 0 (0) | 1 (1)
Weight loss (General disorders) | 0 (0) | 2 (2)
Altered mental status (confusion) (Nervous system disorders) | 0 (0) | 2 (2)
Insomnia (inability to sleep) (Nervous system disorders) | 0 (0) | 1 (1)
Lethargic (Nervous system disorders) | 0 (0) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) — altered blood chemistry affecting the brain
Vertigo (dizziness or syncope) (Nervous system disorders) | 0 (0) | 4 (4)
Difficulty urinating (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (blood in urine) (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chills (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Difficulty of breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Epistaxis (nosebleed) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Fever (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Petechiae (skin spots) (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Pruritus (itching) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No